CLINICAL TRIAL: NCT00868244
Title: Relationship of Facial Pattern With Bruxism
Acronym: BRUXISM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Carlos Martínez Torres, Facultad de medicina de León
Other Study IDs: FMDleoncarlos
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Bruxism
Keywords: facial patterns; bruxism; masticatory muscles
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if the facial pattern is related to the degree of bruxism because the muscles of mastication are the factors of force to the wear of the teeth.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Age 18 to 60 years
3. Case studies to understand orthodontic intraoral photographs of the upper and lower dental arches, and models of lateral skull radiography for orthodontic
4. Cases with any facial biotype development.

Exclusion Criteria:

1. Totally toothless people
2. Partially toothless the posterior (include both molars and premolars).
3. Dawn Syndrome,alzheimer , partial or bilateral facial palsy, autism, which manifest with bruxism
4. Some other syndrome which alters the pattern of facial development as Pierre Robin,crouzon

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: radiographs, photographs and dental plaster models of people who come to orthodontic treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Martinez Torres, León, Guanajuato, Mexico